CLINICAL TRIAL: NCT06306274
Title: Topical Tacrolimus for the Amelioration of Breast Cancer-related Lymphedema: a Randomized, Double-blind, Placebo-controlled Phase II/III Trial
Brief Title: Topical Tacrolimus for Breast Cancer-related Lymphedema
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TACLE trial
Record Dates: First submitted 2024-02-27; First posted 2024-03-12 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: Tacrolimus
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus (0,1%) ointment
  Arms: Active
Drug: Placebo — Placebo ointment
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate the effect of tacrolimus ointment in women with stage I or II breast cancer-related lymphedema. The main question it aims to answer are:

* How tacrolimus affects breast cancer related lymphedema regarding subjective and objective measures (e.g. arm volume, lymphedema index, lymphatic function, and quality of life).
* If maintenance treatment is effective. Participants will be treated with either active drug or placebo once daily for six months followed by a six month maintenance periode with treatment twice weekly. Assessments will be performed at baseline, three, six, nine and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* BCRL ISL stage I or II
* Pitting edema
* Postmenopausal or use of Contraceptive drugs
* Healthy opposite arm
* L-Dex score over 10

Exclusion Criteria:

* Pregnant, breast-feeding, or aiming to conceive within the next year
* Bilateral breast cancer
* Contralateral lymphadenectomy
* Allergy to tacrolimus, macrolides, or iodine
* Pacemaker
* Known kidney or liver disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Lymphedema volume | Baseline to 12 months
  Change in lymphedema volume (volume of lymphedema arm - volume of healty arm)

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Odense University Hospital, Odense
  - Zealand University Hospital, Roskilde
  - Lillebaelt Hospital, Vejle

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hansen FG, Jorgensen MG, Thomsen JB, Sorensen JA. Topical tacrolimus for the amelioration of breast cancer-related lymphedema (TACLE Trial): a study protocol for a randomized, double-blind, placebo-controlled phase II/III trial. Trials. 2025 Apr 8;26(1):127. doi: 10.1186/s13063-025-08829-3. PMID 40200322